CLINICAL TRIAL: NCT07012317
Title: A Randomized, Double-Blind Crossover Trial to Assess Gastrointestinal Responses to Dietary Fibers in Adults Using Weight Loss Medications
Brief Title: A Trial to Assess Gastrointestinal Responses to Dietary Fibers in Adults Using Weight Loss Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2505
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Symptoms; Weight Loss; GLP-1
MeSH Terms: conditions — Weight Loss | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental - Inulin (Experimental)
  Interventions: Other: High Fiber Bar with Inulin
- Experimental - Fiber Blend (Experimental)
  Interventions: Other: High Fiber bar with Fiber Blend
- Experimental - Resistant Starch Type 4 (Experimental)
  Interventions: Other: High Fiber Bar with Resistant Starch type 4
- Control - Low Fiber (Placebo Comparator)
  Interventions: Other: Low Fiber Bar

INTERVENTIONS:
Other: High Fiber Bar with Inulin — Bar with Inulin - high fiber
  Arms: Experimental - Inulin
Other: High Fiber bar with Fiber Blend — Bar with a fiber blend of psyllium husk and bran fibers - high fiber
  Arms: Experimental - Fiber Blend
Other: High Fiber Bar with Resistant Starch type 4 — Bar with Resistant Starch type 4 - High Fiber
  Arms: Experimental - Resistant Starch Type 4
Other: Low Fiber Bar — Snack Bar - Low Fiber
  Arms: Control - Low Fiber

SUMMARY:
The objective of this study is to assess self-reported gastrointestinal (GI) responses to three snack bars containing fiber/fiber blends vs. a control snack bar for 7 days each in adults using GLP-1 agonists.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 25 to 64 years of age, inclusive. There will be approximately equal numbers of men and women.
2. Individual has a self-reported BMI of 18.5 to 39.9 kg/m2, inclusive.
3. Individual has been taking tirzepatide (≥10 mg weekly injection), semaglutide (≥2.0 mg weekly injection), or liraglutide (≥2.4 mg daily injection) for at least 4 weeks and plans to continue to take it throughout the duration of the study.
4. Individual has attained a high school diploma or a General Educational Development (GED) equivalent.
5. Individual has not participated in another research study within 30 days of the screening visit.
6. Individual is willing and able to undergo the scheduled study procedures.
7. Individual understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results. Health conditions may include history or presence of clinically important GI, cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator. Clinically important GI conditions included but are not limited to: inflammatory bowel disease, irritable bowel syndrome, gastroparesis, clinically important lactose intolerance.
2. Individual habitually consumes >8 g fiber per 1000 kcal per day.
3. Individual had a recent (within two weeks of screening) episode of acute GI illness such as nausea, vomiting, or diarrhea.
4. Individual has a history of frequent diarrhea or constipation prior to beginning GLP-1 receptor agonist that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
5. Individual has a history of stomach or GI surgery (e.g., gastric bypass, cholecystectomy) that in the opinion of the Investigator, could interfere with evaluation of the study outcomes.
6. Individual uses medications (over-the counter or prescription) or dietary supplements known to influence gastrointestinal motility including laxatives, enemas, or suppositories; prokinetic drugs; anti-diarrheal agents, anti-spasmotics; fiber supplements; and prebiotic and probiotic supplements (Appendix 6). A 14-day washout phase prior to day 1 is allowed for participants taking any of these products.
7. Daily use of non-steroidal anti-inflammatory drugs (NSAIDs).
8. Individual has a history of cancer in the prior 2 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
9. Individual has a history of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
10. History of any major trauma or major surgical event within 2 months of visit 1.
11. Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1.
12. Use of hemp/marijuana products within 12 months of visit 1. Occasional use (e.g., once or twice a month) within 12 months of visit 1 is allowed but requires at least a 14-day washout prior to day 1 and the participant must be willing to refrain from use during the study.
13. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
14. Individual has an allergy, sensitivity, or intolerance to any foods.
15. Individual has extreme dietary habits (e.g., vegan, Atkins diet, etc.).
16. Individual has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 10 days prior to any visit (washout is permitted for re-scheduling of a visit).
17. Individual has a current or recent history (past 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
18. Individual has been exposed to any non-registered drug product within 30 days prior to screening.
19. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Composite GI Symptom Score | Measured on days 1-10, 25-34, 49-58, and 73-82 where day 1 is the virtual visit date and start of the 3-day baseline. Study product consumption begins on day 4, 28, 52, and 76 and continues for 7 days followed by a 14 day washout period.
  Composite GI Symptom Score is from the GI Tolerability Questionnaire. The composite score will be calculated as the sum of the individual components (nausea, abdominal pain, bloating, intestinal rumbling, and flatulence). The ratings will be coded as: 1 = none/much less than usual, 2 = less than usual, 3 = about usual, 4 = more than usual, and 5 = much more than usual. There will be one composite score per day. Baseline will be defined as the average of the composite scores for the 3-day baseline period. The value for each intervention will be defined as the average of the composite scores for the 7-day intervention period.

SECONDARY OUTCOMES:
Change from baseline in the ratings for the individual component scores of the GIL Tolerability Questionnaire (nausea, abdominal pain, bloating, intestinal rumbling, and flatulence). | Measured on days 1-10, 25-34, 49-58, and 73-82 where day 1 is the virtual visit date and start of the 3-day baseline. Study product consumption begins on day 4, 28, 52, and 76 and continues for 7 days followed by a 14 day washout period.
  For each individual component, the ratings for the 3-day baseline period and the 7-day intervention period will be summed and divided by 3 and 7, respectively, before the change from baseline is calculated.
The frequency of the individual component scores of the GI Tolerability Questionnaire (nausea, abdominal pain, bloating, intestinal rumbling, and flatulence) of 4 or higher (more than usual or much more than usual) during the 7-day intervention period. | Measured on days 1-10, 25-34, 49-58, and 73-82 where day 1 is the virtual visit date and start of the 3-day baseline. Study product consumption begins on day 4, 28, 52, and 76 and continues for 7 days followed by a 14 day washout period.
Change from baseline in the Bristol Stool Form Scale (BSFS) | Measured on days 1-10, 25-34, 49-58, and 73-82 where day 1 is the virtual visit date and start of the 3-day baseline. Study product consumption begins on day 4, 28, 52, and 76 and continues for 7 days followed by a 14 day washout period.
  The scores for the 3-day baseline period and the 7-day intervention period will be summed and divided by the number of bowel movements that occurred during the respective period before the change from baseline is calculated.
Change from baseline in the ratings of stool hardness, straining, discomfort, and incomplete evacuation. | Measured on days 1-10, 25-34, 49-58, and 73-82 where day 1 is the virtual visit date and start of the 3-day baseline. Study product consumption begins on day 4, 28, 52, and 76 and continues for 7 days followed by a 14 day washout period.
  The raitings for the 3-day baseline period and the 7-day intervention period will be summed and divided by the number of bowel movements that occurred during the respective period before the change from baseline is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (2):
- United States (2):
  - Excellence Medical and Research, Miami Gardens, Florida
  - Health Awareness, Port Saint Lucie, Florida